CLINICAL TRIAL: NCT02092935
Title: A Phase II, Randomized, Double-Blind, Active-Controlled Clinical Study to Investigate the Efficacy and Safety of SMT19969 Compared With Vancomycin for the Treatment of Clostridium Difficile-Associated Diarrhoea (CDAD)
Brief Title: A Study of SMT19969 Compared With Vancomycin for the Treatment of Clostridium Difficile-Associated Diarrhoea (CDAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMT19969/C002
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Clostridium Difficile Infection
Keywords: CDAD; Clostridium Difficile
MeSH Terms: conditions — Clostridium Infections | interventions — ridinilazole; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMT19969 (Experimental): 200 mg capsule of SMT19969 twice a day for 10 days with alternating 200 mg placebo twice a day
  Interventions: Drug: SMT19969
- Vancomycin (Active Comparator): 125 mg capsule four times a day for 10 days
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: SMT19969
  Arms: SMT19969
Drug: Vancomycin
  Arms: Vancomycin

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of a new oral antibiotic called SMT19969 in treating C. difficile Infection (CDI).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Clinical diagnosis of CDAD plus laboratory diagnostic test
* No more than 24 hrs antimicrobial treatment for current CDAD episode
* No more than 3 episodes of CDAD in prior 12 months
* No previous episode of CDAD within 30 days of study enrollment
* Female subjects of childbearing potential must use adequate contraception

Exclusion Criteria:

* Life-threatening or fulminant colitis
* Concurrent use of antibiotics or any other treatments for CDAD
* History of inflammatory bowel disease (ulcerative colitis, Crohn's disease)
* Participation in other Clinical research studies within one month of screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the clinical outcome by assessment of sustained clinical response | 30 days post End of Therapy
  Sustained clinical response is defined as clinical cure at the Test of Cure Visit (Day 12) and no recurrence of CDAD within 30 days of End of Therapy

SECONDARY OUTCOMES:
Plasma and faecal concentrations of SMT19969 | 40 Days
  Using laboratory analysis
To assess the safety and tolerability of SMT19969 compared with vancomycin | 40 days
  Assessment of the Adverse Events (AEs) and Serious Adverse Events (SAEs) reported within the study

OTHER OUTCOMES:
To assess the qualitative and quantitative effect of SMT19969 and Vancomycin on the bowel flora of subjects | 40 days
  Using microbiology, sequencing, metagenomic and bioinformatics techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Vickers, PhD, Study Director — Summit (Oxford) Limited
Locations (26):
- United States (24):
  - Mobile, Alabama
  - Laguna Hills, California
  - Long Beach, California
  - Sylmar, California
  - Ventura, California
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Topeka, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Tupelo, Mississippi
  - Billings, Montana
  - Butte, Montana
  - Sommers Point, New Jersey
  - Rochester, New York
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Lima, Ohio
  - Rapid City, South Dakota
  - Seattle, Washington
- Canada (2):
  - Hamilton, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Snydman DR, McDermott LA, Thorpe CM, Chang J, Wick J, Walk ST, Vickers RJ. Antimicrobial susceptibility and ribotypes of Clostridium difficile isolates from a Phase 2 clinical trial of ridinilazole (SMT19969) and vancomycin. J Antimicrob Chemother. 2018 Aug 1;73(8):2078-2084. doi: 10.1093/jac/dky135. PMID 29718329
- [Derived] Vickers RJ, Tillotson GS, Nathan R, Hazan S, Pullman J, Lucasti C, Deck K, Yacyshyn B, Maliakkal B, Pesant Y, Tejura B, Roblin D, Gerding DN, Wilcox MH; CoDIFy study group. Efficacy and safety of ridinilazole compared with vancomycin for the treatment of Clostridium difficile infection: a phase 2, randomised, double-blind, active-controlled, non-inferiority study. Lancet Infect Dis. 2017 Jul;17(7):735-744. doi: 10.1016/S1473-3099(17)30235-9. Epub 2017 Apr 28. PMID 28461207